CLINICAL TRIAL: NCT05694286
Title: A Prospective Evaluation of Infraorbital Filler Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ivona Percec, Principal Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 852212
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-05

CONDITIONS: Dermal Filler; Rejuvenation
Keywords: injectables; tear trough rejuvenation; aesthetic improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infraorbital Filler (Experimental): Receives 1-2mL injection of approved filler in infraorbital region
  Interventions: Procedure: Juvederm Volbella XC hyaluronic acid dermal filler injection

INTERVENTIONS:
Procedure: Juvederm Volbella XC hyaluronic acid dermal filler injection — Infraorbital filler injection

SUMMARY:
The goal of this clinical trial is to measure the facial volumetric changes over time in patients injected with hyaluronic acid dermal filler (Juvéderm Volbella XC) in the infraorbital (under eye) region. Participants will be injected with Juvéderm Volbella XC filler and asked to return for 3D photography at 2 weeks, 1 month, and 3 months post-injection.

DETAILED DESCRIPTION:
Undereye or infraorbital hollowing is a result of a loss of volume causing shadowing and darkness of the infraorbital region often interpreted as a tired, stressed, and aged appearance.

The goal of this clinical trial is to measure the facial volumetric changes over time in patients injected with hyaluronic acid dermal filler (Juvéderm Volbella XC) in the infraorbital (under eye) region. Participants will be injected with Juvéderm Volbella XC filler and asked to return for 3D photography and to complete a validated patient satisfaction questionnaire at 2 weeks, 1 month, and 3 months post-injection. 3D photogrammetry technology allows for high level feature enhancement and microscopic anatomical evaluation that was not previously possible and can be used to make volumetric measurements at injection sites to evaluating minimally invasive injection efficacy.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 22 to 65
* interested in filler injections to reduce undereye volume loss

Exclusion Criteria:

* male
* age <22 or >65
* prior undereye filler
* filler/neurotoxin injection within the past 12 months
* prior facial cosmetic surgery
* prior facial trauma
* planned dental work within next 2 weeks
* travel 1 week prior or 2 weeks after injection

Ages: 22 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivona Percec, MD, PhD, Principal Investigator — Penn Medicine
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infraorbital Filler
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infraorbital Filler
Number analyzed (Participants) | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39.6 [29.9 to 58.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 24.9 [22.0 to 29.1]

OUTCOME MEASURES:

1. Primary Outcome: Volumetric Change in Infraorbital Treatment Baseline to Each Post-intervention Timepoint Day 14, Day 30, and Day 90
Description: 3D facial imaging to measure volumetric changes in the infraorbital region
Time Frame: Post-intervention, Day 14, Day 30, Day 90
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Infraorbital Filler
Number analyzed (Participants) | 11
cc
  Post-injection Day 14 | -0.026 (0.044)
  Post-injection Day 30 | -0.065 (0.054)
  Post-injection Day 90 | -0.108 (0.057)

2. Secondary Outcome: Patient Satisfaction With Validated the Questionnaire FACE-Q
Description: Patient Satisfaction using the validated the questionnaire FACE-Q for patient reported outcomes. Higher scores reflect a better outcome.
Time Frame: Day 0 pre-intervention, Day 0 post-intervention, Day 14, Day 30, Day 90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infraorbital Filler
Number analyzed (Participants) | 11
score on a scale
  FACE-Q - Satisfaction with Eyes at Day 0 pre-injection (minimum score is 0, maximum score is 100) | 46.4 (9.5)
  FACE-Q - Satisfaction with Eyes at Day 0 immediate post-injection (min score is 0, max score is 100) | 59.9 (14.7)
  FACE-Q - Satisfaction with Eyes at Day 14 post-injection (minimum score is 0, maximum score is 100) | 61.4 (13.9)
  FACE-Q - Satisfaction with Eyes at Day 30 post-injection (minimum score is 0, maximum score is 100) | 66.6 (16)
  FACE-Q - Satisfaction with Eyes at Day 90 post-injection (minimum score is 0, maximum score is 100) | 63.4 (19.1)
  FACE-Q - Appraisal of Lower eyelids at Day 0 pre-injection (minimum score is 0, max score is 100) | 55.4 (11.9)
  FACE-Q - Appraisal of Lower eyelids Day 0 immediate post-injection (min score 0, max score is 100) | 65.6 (19.6)
  FACE-Q - Appraisal of Lower eyelids at Day 14 post-injection (minimum score is 0, max score is 100) | 71.1 (13.5)
  FACE-Q - Appraisal of Lower eyelids at Day 30 post-injection (minimum score is 0, max score is 100) | 68.5 (14.1)
  FACE-Q - Appraisal of Lower eyelids at Day 90 post-injection (minimum score is 0, max score is 100) | 66.7 (15.2)
  FACE-Q - Aging Appraisal at Day 0 pre-injection (minimum score is 0, maximum score is 100) | 58.5 (23.9)
  FACE-Q - Aging Appraisal at Day 0 immediate post-injection (minimum score is 0, max score is 100) | 62.5 (25)
  FACE-Q - Aging Appraisal at Day 14 post-injection (minimum score is 0, maximum score is 100) | 60.1 (22.3)
  FACE-Q - Aging Appraisal at Day 30 post-injection (minimum score is 0, maximum score is 100) | 62.6 (18)
  FACE-Q - Aging Appraisal at Day 90 post-injection (minimum score is 0, maximum score is 100) | 64.2 (20.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Infraorbital Filler
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT05694286/Prot_SAP_000.pdf